CLINICAL TRIAL: NCT05616559
Title: The BrainDrugs-Depression Study: A Prospective Precision Psychiatry Cohort Study in the Treatment of Depression
Brief Title: Precision Medicine in the Depression Treatment
Acronym: BDD
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Center for Integrated Molecular Brain Imaging, Copenhagen, Denmak (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Gitte Moos Knudsen, MD,Professor, Rigshospitalet, Denmark
Other Study IDs: H-20083013
Record Dates: First submitted 2022-11-03; First posted 2022-11-15 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorder, Major; Treatment Outcome; Cognitive Dysfunction; Cognitive Behavioral Therapy; Antidepressive Agents
Keywords: PET; MRI; fMRI; EEG; Prediction of treatment response; Early life stress; Selective Serotonin Reuptake Inhibitor; Psychometrics; MDD; Cold cognition; Social cognition; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient cohort (n=800): All participants included will contribute with basic clinical, cognitive, psychometric, genetic and biochemical data.
  Interventions: Combination Product: Treatment Package for First-Episode Depression
- Subcohort I (n=600): Patients in Subcohort I undergo MRI and EEG in addition to expanded clinical, cognitive, psychometric, and biological data.
  Interventions: Combination Product: Treatment Package for First-Episode Depression
- Subcohort II - drug naive PET subgroup (n=60): A subgroup of Subcohort I, including only patients who at inclusion do not receive any pharmacological treatment for their depression, undergo in addition Positron Emission Tomography imaging with [11C]-UCB-J for measurement of cerebral synaptic density.
  Interventions: Combination Product: Treatment Package for First-Episode Depression

INTERVENTIONS:
Combination Product: Treatment Package for First-Episode Depression — The outpatient 'treatment package' for first episode depression is a national uniform package designed by Mental Health Services in the Capital Region. The treatment package for first-episode depression is a program with manualized group CBT, psychoeducation of patients and relatives, and relapse prevention. Antidepressant medication and individual psychotherapy are available as needed.

SUMMARY:
The BrainDrugs-D study uses multimodal neuroimaging combined with self-report measures, clinical and molecular markers to identify clinically relevant predictors that can identify subtypes of major depressive disorder (MDD) and, in a naturalistic setting, predict treatment response to standard antidepressive treatment. The cohorts are followed in nationwide health registries.

DETAILED DESCRIPTION:
BrainDrugs-D is a cohort study of patients with major depressive disorder (MDD) who are deeply phenotyped with demographic, clinical, genetic, biochemical and neuroimaging modalities. These features are subsequently examined for their ability to identify subtypes of MDD and to predict treatment response.

Treatment and study population All participants are phenotyped before initiating a standardized 'treatment package' in out-patient clinics within the Mental Health Services in the Capital Region of Denmark. The goal is to recruit a total of 800 patients with non-psychotic MDD. We use broad inclusion criteria to enable recruitment of representative adult out-patients with non-psychotic MDD who receive standard treatment in practice.

As the study is designed with a high degree of ecological validity, it will not interfere with or delay the standard treatment package for depression. The treatment package is a national uniform package designed by Mental Health Services in the Capital Region, it has been in use since 2017, after several preceding years of clinical use and patient experience. Treatment for first-episode depression has a manualized group Cognitive-behavioural therapy (CBT) as the backbone: 2-3 hours of initial workup followed by 6 hours of individual therapy or 12 sessions of 2 hours of group therapy (8 patients per group), 1-2 hours of engagement and psychoeducation of relatives, 1-5 hours of medication clinic and 2 hours of relapse prevention. Antidepressant medication and individual psychotherapy are instituted, as needed.

Groups The study comprises three groups: The entire cohort (n=800) will have basic clinical, cognitive, psychometric, and biological data available. A subgroup (Subcohort I, n=600) provided expanded clinical, cognitive, psychometric, and biological data as well as Magnetic Resonance Imaging (MRI) and Electroencephalogram (EEG). Subcohort II, (n=60) will be exclusively for patients unmedicated at initiation, consisting of the same investigation, and contributing Positron Emission Tomography imaging with the [11C]-UCB-J tracer of synaptic density.

Follow-up All cohorts receive questionnaires assessing depression symptom severity, level of functioning, and QoL at the three follow-up time points. We also assess the side effects of psychological treatment and medication at the end of the treatment package. The cohorts are also followed in nationwide health registries.

Outcomes The primary outcome is remission (QIDS ≤5) and clinical improvement (≥50% reduction in QIDS) after 6 months.

Secondary endpoints include remission status 12 and 18 months after treatment start and change in QIDS, SCL10, WHO-5, and SDS scores from baseline to follow-ups.

Analysis We will use machine learning algorithms to determine a combination of baseline characteristics that best predict treatment outcomes and statistical models to investigate the association between individual and clinical outcomes. We will also assess associations between patient characteristics, treatment choices, and clinical outcomes using path analysis, enabling us to estimate the effect of treatment choices and timing on the clinical outcome.

Hypotheses for the whole cohort:

Primary hypotheses:

1.1 Clinical, cognitive, psychometric, genetic, and blood biomarker measures at inclusion can predict clinical remission (defined as QIDS≤5) at the first follow-up.

1.2 Clinical, cognitive, psychometric, genetic, and blood biomarker measures at inclusion can predict clinical improvement (a ≥50% reduction in QIDS from pretreatment) at the first follow-up.

Secondary hypotheses:

1.3 Composite scores across a range of clinical, cognitive, psychometric, genetic, and blood biomarker measures at inclusion can cluster patients into MDD subgroups associated with treatment trajectories and outcomes.

1.4 Clinical, cognitive, psychometric, genetic, and blood biomarker measures at inclusion are associated with clinical outcome defined as a change in QIDS.

1.5 Path analysis of baseline patient characteristics and treatment tracks can uncover causal paths for clinical improvements, i.e., estimate the effect of treatment on clinical outcomes.

Hypotheses for Subcohort I

Primary hypotheses:

2.1 MRI, fMRI, and EEG patterns at inclusion may be associated with depressive phenotypes.

2.2 Adding EEG, MRI, and fMRI measures at inclusion to the classifier model (defined in hypotheses 1.1 and 1.2) may significantly improve the prediction of clinical remission and improvement.

Secondary hypotheses:

2.3 Adding EEG, MRI, and fMRI measures at inclusion to the composite score (defined in hypothesis 1.3) may significantly improve the clustering of patients into MDD subgroups.

Hypotheses for Subcohort II

Primary hypotheses:

3.1 Cerebral [11C]-UCB-J binding is lower in patients with MDD than in healthy controls.

3.2 Domain-specific cognitive function correlates positively with [11C]-UCB-J binding in associated cortical and subcortical areas.

Secondary hypotheses:

3.1 Depression severity, anxiety, and anhedonia correlate with [11C]-UCB-J binding in associated cortical and subcortical areas.

3.2 Addition of [11C]-UCB-J binding, EEG, and MRI measures at inclusion to the composite score (defined in hypotheses 2.1) can significantly improve the prediction of clinical improvement and remission beyond clinical, cognitive, psychometric, fluid biomarker, EEG, and MRI measures in antidepressant naïve patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Fulfilment of International Classification of Diseases version 10 diagnostic criteria for a primary depressive episode (i.e., not secondary to known organic or other psychiatric disorder).
* Referral to a treatment package for single-episode depression.

Exclusion Criteria:

* Psychosis or psychotic symptoms
* History of severe head trauma
* Somatic disease associated with morphological brain changes (e.g., brain tumour)
* Insufficient Danish language skills to complete questionnaires and cognitive testing

Additional exclusion criteria for Cohort II:

* Severe somatic disease
* Contraindications for MRI (e.g., metal implants, claustrophobia or back problems)

Additional exclusion criteria for Cohort III:

* Severe somatic disease
* Contraindications for MRI
* Exposure to radioactivity >10 mSv within the last year
* Pregnancy or breastfeeding
* Use of psychotropic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Capital Region of Denmark is the most urban area of Denmark and has a population of 1.6 million people. Patients in the Capital Region of Denmark are referred from their general practitioner or other treatment providers for treatment within the mental health services in the region. All six clinics in the region provide treatment packages for first-episode depression.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Baseline to 6 months after treatment start
  Quick Inventory of Depressive Symptomatology (QIDS) score of ≤5
Clinical improvement | Baseline to 6 months after treatment start
  ≥50% reduction in QIDS score.

SECONDARY OUTCOMES:
Changes in depression severity | Baseline to 6, 12 and 18 months after treatment start
  Changes in depression severity by QIDS (range from 0 to 27, higher score indicating greater severity)
Changes in symptomatology | Baseline to 6, 12 and 18 months after treatment start
  Changes on the Brief Symptom Inventory 18 (BSI-18, range 0-72, higher score indicating greater psychological distress)
Changes in depression and anxiety symptomatology | Baseline to 6, 12 and 18 months after treatment start
  Changes on the 10-item depression and anxiety symptom checklist (SCL-10, range 0-100 higher score indicating greater symptomatology)
Change in wellbeing | Baseline to 6, 12 and 18 months after treatment start
  Changes measured by the WHO-5 well-being Index (range 0-100, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being).
Change in disability | Baseline to 6, 12 and 18 months after treatment start
  Changes measured by modified S. Disability Scale (mSDS) scores (range 0-30, with greater score indicating greater disability)

OTHER OUTCOMES:
Medication side-effects | Baseline to 6 months after treatment start
  Patient Reported Inventory of Side-Effects (PRISE)
Adverse and unwanted events in psychotherapy | Baseline to 6 months after treatment start
  Negative Effects Questionnaire (NEQ) to assess adverse and unwanted events in psychological treatment
Psychosocial remission | Baseline to 6, 12 and 18 months after treatment start
  Defined as either a WHO-5 score of >49, an SCL-10 score of <26 or an mSDS score of <10.

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Jørgensen, DMSc, Principal Investigator — Psychiatric Center Copenhagen; Gitte MK Knudsen, DMSc, Study Director — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via the Center for Integrated Molecular Brain Imaging (Knudsen et al. 2016, NeuroImage), data will be available for the research community upon request and after approval by the scientific board at Neurobiological Research Unit.
  The data will be stored on a password-protected survey system behind secure "firewalls" per the General Data Protection Regulation (GDPR, Regulation European Union (EU) 2016/679 April 27th, 2016) and the Danish Data Protection Act and the regulation (Act No. 502 of May 23rd, 2018). Potential further processing in other national and international laboratories may occur, yet always per the GDPR (Regulation EU 2016/679 April 27th, 2016), the Danish Data Protection Act, and the regulation (Act No. 502 of May 23rd, 2018).
Time Frame: Upon study completion
Access Criteria: Researchers may apply for access to the data.
URL: https://nru.dk/index.php/research-menu/research-groups/115-the-cimbi-database-and-biobank

REFERENCES:
- [Background] Cipriani A, Furukawa TA, Salanti G, Chaimani A, Atkinson LZ, Ogawa Y, Leucht S, Ruhe HG, Turner EH, Higgins JPT, Egger M, Takeshima N, Hayasaka Y, Imai H, Shinohara K, Tajika A, Ioannidis JPA, Geddes JR. Comparative efficacy and acceptability of 21 antidepressant drugs for the acute treatment of adults with major depressive disorder: a systematic review and network meta-analysis. Lancet. 2018 Apr 7;391(10128):1357-1366. doi: 10.1016/S0140-6736(17)32802-7. Epub 2018 Feb 21. PMID 29477251
- [Background] Trevino K, McClintock SM, McDonald Fischer N, Vora A, Husain MM. Defining treatment-resistant depression: a comprehensive review of the literature. Ann Clin Psychiatry. 2014 Aug;26(3):222-32. PMID 25166485
- [Background] Kessler RC, van Loo HM, Wardenaar KJ, Bossarte RM, Brenner LA, Ebert DD, de Jonge P, Nierenberg AA, Rosellini AJ, Sampson NA, Schoevers RA, Wilcox MA, Zaslavsky AM. Using patient self-reports to study heterogeneity of treatment effects in major depressive disorder. Epidemiol Psychiatr Sci. 2017 Feb;26(1):22-36. doi: 10.1017/S2045796016000020. Epub 2016 Jan 26. PMID 26810628
- [Derived] Jensen KHR, Dam VH, Ganz M, Fisher PM, Ip CT, Sankar A, Marstrand-Joergensen MR, Ozenne B, Osler M, Penninx BWJH, Pinborg LH, Frokjaer VG, Knudsen GM, Jorgensen MB. Deep phenotyping towards precision psychiatry of first-episode depression - the Brain Drugs-Depression cohort. BMC Psychiatry. 2023 Mar 9;23(1):151. doi: 10.1186/s12888-023-04618-x. PMID 36894940
- See also: Description of treatment package (in Danish) — https://www.regioner.dk/media/11322/pakkeforloeb-for-depressiv-enkelt-episode.pdf